CLINICAL TRIAL: NCT03048916
Title: Acute Stroke Patients With Dysphagia After Different Swallowing Therapies: Videofluoroscopy Findings and Brain Plasticity in Magnetic Resonance Imaging
Brief Title: Dysphagia After Different Swallowing Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMRPG896021
Record Dates: First submitted 2017-02-05; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Dysphagia; Videofluoroscopy; Stroke
Keywords: dysphagia; stroke; magnetic resonance imaging; videofluoroscopy
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- general swallowing therapy (Other): including:
  * oral exercises
  * tactile stimulation
  * compensatory techniques
  * swallowing maneuvers
  Interventions: Other: general swallowing therapy
- the NMES therapy with VitalStim therapeutic device (Experimental): The placement of 2-channel electrodes is depended on the dysphagic types and the findings on VFS
  Interventions: Other: NMES therapy
- : the combined NMES and general swallowing therapies (Active Comparator)
  Interventions: Other: general swallowing therapy; Other: NMES therapy

INTERVENTIONS:
Other: general swallowing therapy — including a session of oral exercises, tactile stimulation, compensatory techniques, swallowing maneuvers that are taught to the participants by a speech therapist.
  Arms: : the combined NMES and general swallowing therapies; general swallowing therapy
Other: NMES therapy — he NMES therapy with VitalStim therapeutic device will be done by one physician who is licensed practitioner and certified in use of the VitalStim device. The placement of 2-channel electrodes is depended on the dysphagic types and the findings on VFS.
  Arms: : the combined NMES and general swallowing therapies; the NMES therapy with VitalStim therapeutic device

SUMMARY:
Dysphagia after stroke is associated to increased pulmonary complications and mortality. The swallowing therapies could decrease the pulmonary complications and improve the quality of life after stroke. The swallowing therapies include dietary modifications, thermal stimulation, compensatory positions, and oropharyngeal muscle stimulation. Most researchers used clinical assessments and videofluoroscopy to evaluate the effect of the swallowing therapies. Some authors performed functional magnetic resonance imaging (fMRI) to investigate the brain neuroactivity during swallowing with tasks in normal adults and unilateral hemispheric stroke patients. The aim of this study is to explore the effect of swallowing therapies not only in clinical swallowing function but also brain plasticity of acute stroke patients with dysphagia by videofluoroscopy and fMRI.

DETAILED DESCRIPTION:
In the study, 10 healthy controls and 48 patients with a single and acute hemispheric or brain stem stroke will be enrolled. Both 24 hemispheric and 24 brain stem stroke patients will be divided into 3 groups. General swallowing therapy, oropharyngeal neuromuscular electrical stimulation (NMES), and combined general and NMES therapies will be randomly provided for the 3 groups. Each patient will receive clinical assessment of food oral intake scale, functional dysphagia scale of videofluoroscopy, and brain neuroactivity in fMRI.

The investigators hope to find the benefit of the swallowing therapies both in clinical swallowing function and in brain functional neuroactivity/reorganization after acute stroke. While comparing the 3 swallowing therapies, different functional neuroactivity may be facilitated by different swallowing therapies. Finally, the investigators could also find out the most effective swallowing therapy among the 3 therapies in acute stroke patients with dysphagia according to the findings of videofluoroscopy and fMRI.

ELIGIBILITY:
Inclusion criteria of normal controls:

* normal neurological examination
* no history of stroke
* no active neurological disorder

Inclusion criteria of hemispheric stroke patients:

* a single cerebral hemispheric stroke
* swallowing difficulty: detected by bedside swallow assessment by a physician while admitting to the rehabilitation unit.

Inclusion criteria of these brain stem stroke patients:

* a single brain stem stroke without prior stroke history
* swallowing difficulties: detected by bedside swallow assessment by a physician while admitting to the rehabilitation unit

Exclusion criteria:

* multiple brain lesions due to one episode of stroke
* impaired communication ability due to cognition deficit
* other central or peripheral neurological deficit leading to swallowing difficulty.
* use of an electrically sensitive biomedical device (eg. cardiac pacemaker)
* metal clip in the brain
* pneumonia at the time of enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2013-07-31 (Actual)

PRIMARY OUTCOMES:
The functional oral intake scale | baseline (before intervention), changes from baseline FOIS at 4 weeks
  Clinical swallowing evaluations: The functional oral intake scale (FOIS) was reported by Crary et al. for presenting the functional oral intake of food and liquid in stroke patients. One physician who is blinded to the therapies will evaluate the FOIS for each participant before and after swallowing treatments.

SECONDARY OUTCOMES:
8-point penetration-aspiration scale (PAS) | baseline (before intervention), changes from baseline PAS score at 4 weeks
  VFS is a standard tool for swallowing disorders. A 8-point penetration-aspiration scale (PAS) is used for observing the event of penetration or aspiration on VFS.
11-item functional dysphagia scale (FDS) | baseline (before intervention), changes from baseline FDS score at 4weeks
  A 11-item functional dysphagia scale (FDS) of VFS is a sensitive and specific method for quantifying swallowing function in stroke.
3-Dimensional (3D) structural MRI | baseline (before intervention), changes from baseline result of 3-Dimensional (3D) structural MRI at 4 weeks
  MR images are obtained using a 3.0-T whole body magnet with a 50- and 23-mT/m gradient strength, and an echo-planar-capable receiver (GE SIGNA EXCITE HD, GE Medical Systems, Milwaukee, US).
  A 3-dimensional (3D) structural MRI is acquired for each subject using a T1-weighted gradient echo magnetization prepared rapid gradient echo sequence yielding 124 sagittal slices with a defined voxel size of 1 x 1 x 1.5 mm.
Function MRI | baseline (before intervention), changes from baseline result of fMRI at 4 weeks
  MR images are obtained using a 3.0-T whole body magnet with a 50- and 23-mT/m gradient strength, and an echo-planar-capable receiver (GE SIGNA EXCITE HD, GE Medical Systems, Milwaukee, US).
  The functional images are obtained using an EPI sequence with the following parameters: 33 axial slices, image resolution = 3.75*3.75*4, and TR= 2000 ms.
Diffusion tensor imaging | baseline (before intervention), changes from baseline result of diffusion tensor imaging at 4 weeks
  MR images are obtained using a 3.0-T whole body magnet with a 50- and 23-mT/m gradient strength, and an echo-planar-capable receiver (GE SIGNA EXCITE HD, GE Medical Systems, Milwaukee, US).
  An 8 channels diffusion tensor imaging (DTI) acquisition protocol will be used to acquire high resolution DTI, i.e. 2 x 2 x 2 mm3 voxel size. With 13 diffusion encoding directions and number of average of 4, whole brain DTI and high resolution eigenvector field can be acquired within 20 mins.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chi Huang, Bachelor, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barer DH. The natural history and functional consequences of dysphagia after hemispheric stroke. J Neurol Neurosurg Psychiatry. 1989 Feb;52(2):236-41. doi: 10.1136/jnnp.52.2.236. PMID 2564884
- [Background] Meng NH, Wang TG, Lien IN. Dysphagia in patients with brainstem stroke: incidence and outcome. Am J Phys Med Rehabil. 2000 Mar-Apr;79(2):170-5. doi: 10.1097/00002060-200003000-00010. PMID 10744192
- [Background] Paciaroni M, Mazzotta G, Corea F, Caso V, Venti M, Milia P, Silvestrelli G, Palmerini F, Parnetti L, Gallai V. Dysphagia following Stroke. Eur Neurol. 2004;51(3):162-7. doi: 10.1159/000077663. Epub 2004 Apr 1. PMID 15073441
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Foley N, Teasell R, Salter K, Kruger E, Martino R. Dysphagia treatment post stroke: a systematic review of randomised controlled trials. Age Ageing. 2008 May;37(3):258-64. doi: 10.1093/ageing/afn064. PMID 18456790
- [Background] Smithard DG, Smeeton NC, Wolfe CD. Long-term outcome after stroke: does dysphagia matter? Age Ageing. 2007 Jan;36(1):90-4. doi: 10.1093/ageing/afl149. Epub 2006 Dec 15. PMID 17172601
- [Background] Goulding R, Bakheit AM. Evaluation of the benefits of monitoring fluid thickness in the dietary management of dysphagic stroke patients. Clin Rehabil. 2000 Apr;14(2):119-24. doi: 10.1191/026921500667340586. PMID 10763787
- [Background] Carnaby G, Hankey GJ, Pizzi J. Behavioural intervention for dysphagia in acute stroke: a randomised controlled trial. Lancet Neurol. 2006 Jan;5(1):31-7. doi: 10.1016/S1474-4422(05)70252-0. PMID 16361020
- [Background] DePippo KL, Holas MA, Reding MJ, Mandel FS, Lesser ML. Dysphagia therapy following stroke: a controlled trial. Neurology. 1994 Sep;44(9):1655-60. doi: 10.1212/wnl.44.9.1655. PMID 7936292
- [Background] Dennis MS, Lewis SC, Warlow C; FOOD Trial Collaboration. Effect of timing and method of enteral tube feeding for dysphagic stroke patients (FOOD): a multicentre randomised controlled trial. Lancet. 2005 Feb 26-Mar 4;365(9461):764-72. doi: 10.1016/S0140-6736(05)17983-5. PMID 15733717
- [Background] Hamidon BB, Abdullah SA, Zawawi MF, Sukumar N, Aminuddin A, Raymond AA. A prospective comparison of percutaneous endoscopic gastrostomy and nasogastric tube feeding in patients with acute dysphagic stroke. Med J Malaysia. 2006 Mar;61(1):59-66. PMID 16708735
- [Background] Burnett TA, Mann EA, Cornell SA, Ludlow CL. Laryngeal elevation achieved by neuromuscular stimulation at rest. J Appl Physiol (1985). 2003 Jan;94(1):128-34. doi: 10.1152/japplphysiol.00406.2002. PMID 12486019
- [Background] Park CL, O'Neill PA, Martin DF. A pilot exploratory study of oral electrical stimulation on swallow function following stroke: an innovative technique. Dysphagia. 1997 Summer;12(3):161-6. doi: 10.1007/PL00009531. PMID 9190102
- [Background] Freed ML, Freed L, Chatburn RL, Christian M. Electrical stimulation for swallowing disorders caused by stroke. Respir Care. 2001 May;46(5):466-74. PMID 11309186
- [Background] Leelamanit V, Limsakul C, Geater A. Synchronized electrical stimulation in treating pharyngeal dysphagia. Laryngoscope. 2002 Dec;112(12):2204-10. doi: 10.1097/00005537-200212000-00015. PMID 12461342
- [Background] Ludlow CL, Bielamowicz S, Daniels Rosenberg M, Ambalavanar R, Rossini K, Gillespie M, Hampshire V, Testerman R, Erickson D, Carraro U. Chronic intermittent stimulation of the thyroarytenoid muscle maintains dynamic control of glottal adduction. Muscle Nerve. 2000 Jan;23(1):44-57. doi: 10.1002/(sici)1097-4598(200001)23:13.0.co;2-e. PMID 10590405
- [Background] Hagg M, Larsson B. Effects of motor and sensory stimulation in stroke patients with long-lasting dysphagia. Dysphagia. 2004 Fall;19(4):219-30. doi: 10.1007/s00455-004-0016-3. PMID 15667056
- [Background] Martin RE, Sessle BJ. The role of the cerebral cortex in swallowing. Dysphagia. 1993;8(3):195-202. doi: 10.1007/BF01354538. PMID 8359039
- [Background] Hamdy S, Rothwell JC, Aziz Q, Thompson DG. Organization and reorganization of human swallowing motor cortex: implications for recovery after stroke. Clin Sci (Lond). 2000 Aug;99(2):151-7. PMID 10918049
- [Background] Ertekin C, Aydogdu I. Neurophysiology of swallowing. Clin Neurophysiol. 2003 Dec;114(12):2226-44. doi: 10.1016/s1388-2457(03)00237-2. PMID 14652082
- [Background] Hamdy S, Aziz Q, Rothwell JC, Crone R, Hughes D, Tallis RC, Thompson DG. Explaining oropharyngeal dysphagia after unilateral hemispheric stroke. Lancet. 1997 Sep 6;350(9079):686-92. doi: 10.1016/S0140-6736(97)02068-0. PMID 9291902
- [Background] Hamdy S, Aziz Q, Rothwell JC, Power M, Singh KD, Nicholson DA, Tallis RC, Thompson DG. Recovery of swallowing after dysphagic stroke relates to functional reorganization in the intact motor cortex. Gastroenterology. 1998 Nov;115(5):1104-12. doi: 10.1016/s0016-5085(98)70081-2. PMID 9797365
- [Background] Hamdy S, Aziz Q, Rothwell JC, Singh KD, Barlow J, Hughes DG, Tallis RC, Thompson DG. The cortical topography of human swallowing musculature in health and disease. Nat Med. 1996 Nov;2(11):1217-24. doi: 10.1038/nm1196-1217. PMID 8898748
- [Background] Hamdy S, Rothwell JC, Aziz Q, Singh KD, Thompson DG. Long-term reorganization of human motor cortex driven by short-term sensory stimulation. Nat Neurosci. 1998 May;1(1):64-8. doi: 10.1038/264. PMID 10195111
- [Background] Robbins J, Levin RL. Swallowing after unilateral stroke of the cerebral cortex: preliminary experience. Dysphagia. 1988;3(1):11-7. doi: 10.1007/BF02406275. No abstract available. PMID 3248391
- [Background] Li S, Luo C, Yu B, Yan B, Gong Q, He C, He L, Huang X, Yao D, Lui S, Tang H, Chen Q, Zeng Y, Zhou D. Functional magnetic resonance imaging study on dysphagia after unilateral hemispheric stroke: a preliminary study. J Neurol Neurosurg Psychiatry. 2009 Dec;80(12):1320-9. doi: 10.1136/jnnp.2009.176214. Epub 2009 Jun 9. PMID 19515639
- [Background] Robbins J, Levine RL, Maser A, Rosenbek JC, Kempster GB. Swallowing after unilateral stroke of the cerebral cortex. Arch Phys Med Rehabil. 1993 Dec;74(12):1295-300. doi: 10.1016/0003-9993(93)90082-l. PMID 8259895
- [Background] Hamdy S, Mikulis DJ, Crawley A, Xue S, Lau H, Henry S, Diamant NE. Cortical activation during human volitional swallowing: an event-related fMRI study. Am J Physiol. 1999 Jul;277(1):G219-25. doi: 10.1152/ajpgi.1999.277.1.G219. PMID 10409170
- [Background] Mosier K, Patel R, Liu WC, Kalnin A, Maldjian J, Baredes S. Cortical representation of swallowing in normal adults: functional implications. Laryngoscope. 1999 Sep;109(9):1417-23. doi: 10.1097/00005537-199909000-00011. PMID 10499047
- [Background] Mosier KM, Liu WC, Maldjian JA, Shah R, Modi B. Lateralization of cortical function in swallowing: a functional MR imaging study. AJNR Am J Neuroradiol. 1999 Sep;20(8):1520-6. PMID 10512240
- [Background] Kern MK, Jaradeh S, Arndorfer RC, Shaker R. Cerebral cortical representation of reflexive and volitional swallowing in humans. Am J Physiol Gastrointest Liver Physiol. 2001 Mar;280(3):G354-60. doi: 10.1152/ajpgi.2001.280.3.G354. PMID 11171617
- [Background] Martin RE, Goodyear BG, Gati JS, Menon RS. Cerebral cortical representation of automatic and volitional swallowing in humans. J Neurophysiol. 2001 Feb;85(2):938-50. doi: 10.1152/jn.2001.85.2.938. PMID 11160524
- [Background] O'Donoghue S, Bagnall A. Videofluoroscopic evaluation in the assessment of swallowing disorders in paediatric and adult populations. Folia Phoniatr Logop. 1999 Jul-Oct;51(4-5):158-71. doi: 10.1159/000021494. PMID 10450023
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Background] Han TR, Paik NJ, Park JW. Quantifying swallowing function after stroke: A functional dysphagia scale based on videofluoroscopic studies. Arch Phys Med Rehabil. 2001 May;82(5):677-82. doi: 10.1053/apmr.2001.21939. PMID 11346847